CLINICAL TRIAL: NCT07181018
Title: Multimorbidity in Metabolic Syndrome: A Longitudinal Cohort Study in TWINS.PL
Brief Title: Metabolic Syndrome Among Polish Twins
Acronym: TWINSPL
Status: Recruiting | Type: Observational
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/ABM/03/00048
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Twins; Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Trial within cohort (TWIC) — Educational intervention based on a protocol specifically developed for the TWINS.PL cohort, aimed at activating and engaging the participant in the intervention process.
  Intervention group: Phenotypically concordant participants from the TWINS.PL STUDY cohort, randomized to receive an educational intervention designed to actively engage them in modifying selected health-relevant endpoints.
  Control group: The co-twin of the participant randomized to the intervention arm, serving as the control.
  1. TWINS-TWIC HL: Research Question: Does participation in a structured, participant-activating educational intervention program influence health literacy indicators among participants of the TWINS.PL study? Study Design: A randomized controlled trial embedded within a prospective observational twin cohort (TWiC study in a twin cohort).
  2. TWINS-TWIC DIET Research Question: Does participation in a structured, participant-activating educational intervention focused on dietary habits influence the

SUMMARY:
Over a 5-year follow-up period, we aim to conduct a study among twins aged 15-44 years from the Polish population with the following objectives:

1. To determine the incidence and risk factors for the development of de novo metabolic dysfunction-associated steatotic liver disease (MASLD), liver fibrosis, or cirrhosis. We also intend to evaluate the progression of hepatic steatosis from early to advanced stages or toward fibrosis/cirrhosis.
2. To determine the prevalence and identify predictive factors for the onset and progression of features, diseases, or complications of metabolic syndrome (MS) other than liver disease, particularly within the spectrum of metabolic, nutritional, cardiovascular, endocrine, oncological, psychological, and other disorders typically associated with MS.
3. To assess the association between previous COVID-19 infection or long-COVID features and the occurrence of MASLD, liver fibrosis, or cirrhosis due to MASLD, as well as other features, diseases, or complications of MS.
4. To evaluate the prevalence of malignancies in a young twin population (aged 15-44 years) with MS or with risk factors for MS.
5. To investigate the contribution of genetic and environmental factors and gut microbiota composition to the development and progression of structural liver changes (steatosis, fibrosis, cirrhosis) in MASLD, as well as other features and complications of MS in twins discordant for the MS phenotype.
6. To assess the role of genetic and environmental components in the occurrence and severity of MS phenotype discordance in monozygotic twins.

ELIGIBILITY:
Inclusion Criteria

1. Age between 15 and 44 years. 2. Provision of informed consent to participate in the study. 3. Twin with a living co-twin. 4. Positive family history in first- and second-degree relatives of metabolic syndrome (MS), associated diseases, or the most common complications of the syndrome.

________________________________________ Exclusion Criteria

Permanent exclusion criteria:

1. Co-twin does not consent to participate in the study.
2. Inability to obtain medical history of biological family members.
3. Presence of advanced liver fibrosis, cirrhosis, or liver cancer.
4. Known liver genetic disorders, autoimmune hepatitis, celiac disease, hemochromatosis, primary biliary cholangitis (PBC), primary sclerosing cholangitis (PSC), cystic fibrosis, or Wilson's disease.
5. Current or chronic alcohol consumption >20 g of ethanol/day in women and >30 g/day in men.
6. Short bowel syndrome.
7. Cyanotic congenital heart defect.
8. Myasthenia.
9. Central nervous system degenerative diseases such as Alzheimer's disease, Parkinson's disease, or Huntington's disease.
10. Storage diseases involving the liver.
11. Active malignant neoplasm undergoing treatment (excluding non-melanoma skin cancers and melanoma treated non-pharmacologically).
12. Chronic kidney disease requiring renal replacement therapy.
13. Status post organ or tissue transplantation requiring immunosuppression.
14. Pituitary, hypothalamic, or adrenal hyperfunction/hypofunction requiring hormone supplementation.
15. Addiction to psychoactive substances or drugs.
16. Other severe and incurable diseases that, in the investigator's opinion, constitute a permanent contraindication for participation in the study.
17. Lack of cooperation by the volunteer during the visit to the Research Center. ________________________________________

Temporary exclusion criteria (after resolution, the volunteer may be enrolled):

1. Acute infection, low-grade fever or fever, or use of antibiotics at the time of recruitment or prior to the visit at the Research Center - inclusion possible after 6 weeks.
2. Any vaccination within the past 6 weeks.
3. Pregnancy and up to 6 months postpartum.
4. 3 months after the natural cessation of breastfeeding.
5. 3 months after surgery (does not apply to minor surgical procedures).
6. Untreated hyperthyroidism or hypothyroidism - inclusion possible 3 months after achieving euthyroidism.
7. Significant weight loss or gain in the past 3 months (>10% of initial body weight) - inclusion possible 3 months after weight stabilization.
8. 6 months after discontinuation of temporary parenteral or enteral nutrition via feeding tube.
9. 12 months after bariatric surgery.
10. Systemic treatment with steroids, chemotherapy, immunosuppressive drugs, or biological therapy known to be hepatotoxic or potentially inducing abnormalities found in MS - inclusion possible at least 3 months after completing therapy.

Ages: 15 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population comprises Polish twin individuals aged 15-44 years, who have provided informed consent, have a living co-twin, and present a positive family history (first- or second-degree relatives) of metabolic syndrome, its related comorbidities, or common complications.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2033-09-30 (Estimated)

PRIMARY OUTCOMES:
De novo occurrence of metabolic steatosis, hepatic fibrosis, or cirrhosis. | Baseline up to approximately 5 years
  De novo occurrence of metabolic steatosis, hepatic fibrosis, or cirrhosis based on assessment by magnetic resonance imaging-proton density fat fraction (MRI-PDFF) and/or transient elastography.
Progression of hepatic steatosis or fibrosis to more advanced stages or cirrhosis. | Baseline up to approximately 5 years
  Progression of hepatic steatosis or fibrosis to more advanced stages or cirrhosis, as assessed by magnetic resonance imaging and dynamic elastography, using the following evaluation scales:
  * The hepatic steatosis grading scale based on magnetic resonance imaging-proton density fat fraction (MRI-PDFF);
  * The hepatic steatosis grading scale based on dynamic elastography using the Controlled Attenuation Parameter (CAP) technique;
  * The liver fibrosis grading scale assessed by dynamic elastography using liver stiffness (LS) measurement, according to the METAVIR scoring system

SECONDARY OUTCOMES:
First-time occurrence of overweight or obesity | Baseline to approximately 5 years
  Overweight will be defined as a BMI of 25 to <30 kg/m², and obesity as a BMI of ≥30 kg/m²
First-time occurrence of an increase in visceral adipose tissue | Baseline to approximately 5 years
  Increase in visceral adipose tissue >10%, as assessed by DEXA or BIA
First-time occurrence of Prediabetes or type 2 diabetes mellitus (T2DM) | Baseline to approximately 5 years
  First diagnosis of prediabetes or type 2 diabetes mellitus (T2DM), confirmed by standard laboratory criteria (fasting plasma glucose, HbA1c, or oral glucose tolerance test) in accordance with current ADA/EASD guidelines
The assessment of HOMA-IR | Baseline to approximately 5 years
  First-time occurrence of HOMA-IR >5
First-time occurrence of Pancreatic steatosis | Baseline to approximately 5 years
  Visualization of pancreatic steatosis during abdominal ultrasound and/or MRI-PDFF
First-time occurrence of Hypertension (HTN) | Baseline to approximately 5 years
  Diagnosis of arterial hypertension according to the ESC/ESH definition
First-time occurrence of Acute coronary syndrome, the need for coronary artery bypass grafting (CABG), any percutaneous coronary intervention (PCI), or detection of regional wall motion abnormalities on echocardiography | Baseline to approximately 5 years
  All outcome events will be confirmed through review of medical records, including hospitalization reports, procedural documentation, and echocardiographic findings, in accordance with the most recent ESC guidelines on Acute Coronary Syndromes.
First-time occurrence of Systolic heart failure with a reduced left ventricular ejection fraction of less than 45% | Baseline to approximately 5 years
  Diagnosis of systolic heart failure confirmed by echocardiographic assessment showing a left ventricular ejection fraction (LVEF) <45%.
First-time occurrence of Atrial fibrillation/flutter | Baseline to approximately 5 years
  First documented episode of atrial fibrillation (paroxysmal, persistent, or permanent) or atrial flutter, confirmed by ECG or other cardiac monitoring, or the need for pulmonary vein isolation and/or cavotricuspid isthmus ablation.
First-time occurrence of Requirement for angioplasty, stenting, or surgery of the aorta or any other arteries (excluding trauma-related causes) | Baseline to approximately 5 years
  First requirement for angioplasty, stent placement, or surgical intervention of the aorta or other arteries (excluding trauma-related procedures), confirmed by medical records and procedural documentation.
First-time occurrence of Implantation of a cardiac electronic device | Baseline to approximately 5 years
  First implantation of a cardiac electronic device (e.g., pacemaker, ICD, or CRT) indicated for sick sinus syndrome, advanced atrioventricular conduction abnormalities, or ischemic heart disease, as confirmed by procedural documentation.
First-time occurrence of Transient ischemic attack (TIA) or ischemic stroke | Baseline to approximately 5 years
  First documented occurrence of transient ischemic attack (TIA) or ischemic stroke, confirmed by neurological assessment and/or neuroimaging, in accordance with current ESC guidelines.
First-time occurrence of Hashimoto's thyroiditis | Baseline to approximately 5 years
  Increase of at least one anti-thyroid autoantibody - anti-thyroid peroxidase and/or anti-thyroglobulin, accompanied by typical ultrasound picture suggesting Hashimoto's thyroiditis, namely irregular, decreased echogenicity of thyroid parenchyma, signs of fibrosis and decreased vascularity on Color Doppler examination
First-time occurrence of Focal thyroid lesions detected on ultrasound | Baseline to approximately 5 years
  Focal thyroid lesions detected on ultrasound (≥1 lesion with a diameter >5 mm)
First-time occurrence of Adrenal incidentaloma | Baseline to approximately 5 years
  Adrenal lesion >10 mm in diameter
First-time occurrence of Malignancy with a known potential association with insulin resistance | Baseline to approximately 5 years
  e.g., colorectal, thyroid, breast, endometrial, hepatic, pancreatic, renal, gallbladder, esophageal, or ovarian cancer
First-time occurrence of Long COVID-19 syndrome | Baseline to approximately 5 years
  Defined as persistent (over 12 weeks) symptoms (listed in the questionnaire filled out by the patient), which appeared after COVID-19 infection and their occurrence cannot be explained by other causes
Death from non-accidental causes | Baseline to approximately 5 years
  The number of deaths from non accidental causes during the observation period
The assessment of HbA1c | Baseline to approximately 5 years
  First-time occurrence of HbA1c >5.7%

CONTACTS AND LOCATIONS:
Locations (1):
- Uniwersytecki Szpital Kliniczny, Poznan, Wielkopolska, Poland

IPD SHARING:
Plan to Share IPD: No